CLINICAL TRIAL: NCT01985256
Title: A Phase 1 Ascending Dose Trial of the Safety and Tolerability of Toca 511, a Retroviral Replicating Vector, Administered Intravenously Prior to, and Intracranially at the Time of, Subsequent Resection for Recurrent HGG & Followed by Treatment With Extended-Release 5-FC
Brief Title: Study of a Retroviral Replicating Vector Given Intravenously to Patients Undergoing Surgery for Recurrent Brain Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tocagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tg 511-13-01
Record Dates: First submitted 2013-11-08; First posted 2013-11-15 (Estimated); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Glioblastoma Multiforme; Anaplastic Astrocytoma; Anaplastic Oligodendroglioma; Anaplastic Oligoastrocytoma
Keywords: glioma; glioblastoma; glioblastoma multiforme; Grade IV astrocytoma; brain cancer; recurrent glioblastoma; GBM; AA; AOD; anaplastic astrocytoma; anaplastic oligodendroglioma; anaplastic oligoastrocytoma; malignant glioma; high grade glioma
MeSH Terms: conditions — Glioblastoma; Astrocytoma; Oligodendroglioma; Glioma; Brain Neoplasms | interventions — vocimagene amiretrorepvec; Flucytosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Experimental): Toca 511 vector/Toca FC
  Interventions: Biological: Toca 511; Drug: Toca FC

INTERVENTIONS:
Biological: Toca 511 — All patients will receive Toca 511, a retroviral replicating vector that expresses the cytosine deaminase (CD) gene, intravenously and then intracranially. CD converts the antifungal 5-fluorocytosine (5-FC) to the anti-cancer drug 5-fluorouracil (5-FU) in cells that have been infected by the Toca 511 vector. Beginning approximately 6 weeks after the second administration of Toca 511,patients will begin 7-day course of oral 5-FC, repeated every 4 weeks for the duration of the study.
  Other Names: vocimagene amiretrorepvec; retroviral replicating vector (RRV)
Drug: Toca FC
  Other Names: flucytosine, 5-FC, 5-FC XR, Toca FC

SUMMARY:
This is a multicenter study evaluating the safety and tolerability of Toca 511 administered intravenously to patients with recurrent or progressive Grade III or Grade IV Gliomas who have elected to undergo surgical removal of their tumor. Patients meeting all of the inclusion and none of the exclusion criteria will receive an initial dose of Toca 511 administered as an intravenous, bolus injection, followed approximately 11 days later by an additional dose injected into the walls of the resection cavity at the time of planned tumor resection. Approximately 6 weeks later, patients will begin treatment with oral Toca FC, an antifungal agent, and repeated every 4 weeks. All patients enrolled in this study will be encouraged to participate in a continuation protocol that enables additional Toca FC administration and the collection of long-term safety and response data.

ELIGIBILITY:
Inclusion Criteria:

* Has the subject given written informed consent?
* Is the subject between 18 years old and 80 years old inclusive?
* Has the subject had histologically proven HGG with recurrence or progression following initial definitive therapy(s) such as surgery with or without adjuvant radiation therapy and/or chemotherapy (confirmed by diagnostic biopsy or contrast-enhanced MRI and evaluable by Macdonald criteria)? Note, if first recurrence of HGG is documented by MRI, an interval of at least 12 weeks after the end of prior radiation therapy is required unless there is either: i) histopathologic confirmation of recurrent tumor, or ii) new enhancement on MRI outside of the radiotherapy treatment field.
* Does the patient have either (1) a single, enhancing tumor recurrence/progression that is ≤ 8 cm in greatest dimension, or (2) multiple enhancing tumor recurrences/progressions within the same surgical field where the sum of their greatest dimensions is ≤ 8 cm?
* Based on the pre-operative evaluation, is the tumor recurrence/progression a candidate for ≥ 80% resection?
* Has the subject elected not to undergo treatment with the Gliadel® wafer?
* Does the subject have a Karnofsky performance status ≥ 70?
* Does the subject have an absolute neutrophil count (ANC) ≥ 1500/mm3?
* Does the subject have an absolute lymphocyte count ≥ 500/mm3?
* Does the subject have a platelet count ≥ 100,000/mm3?
* Does the subject have a Hgb ≥ 10 g/dL?
* Does the subject have a coagulation profile that would allow for the safe performance of surgery under general anesthesia?
* Does the subject have an estimated glomerular filtration rate of at least 50 mL/min (inclusive) by the Cockcroft-Gault formula?
* Does the subject have an ALT < 3 times the upper limit of the laboratory reference range and total bilirubin < 1.5 mg/dL?
* If the subject is a female of childbearing potential, has she had a negative serum pregnancy test within the past 21 days?
* Is the subject willing to use condoms for contraception for 6 months after receiving Toca 511 or until there is no evidence of the virus in his/her blood, whichever is longer. If the subject is a fertile female, is she willing to use contraception for at least 12 months?
* Is the subject willing and able to abide by the protocol?
* Does the subject have adequate venous access?

Exclusion Criteria:

* Has the subject received cytotoxic chemotherapy within the past 3 weeks (6 weeks for nitrosoureas) of the planned date of vector injection?
* Does the subject have, or has the subject had, within the past 4 weeks any infection requiring antibiotic, antifungal or antiviral therapy?
* Has the subject received Avastin® (bevacizumab) for this recurrence/progression, or within the 4 weeks prior to planned Visit 1?
* Does the subject have any bleeding diathesis, or must the subject take any anticoagulants, or antiplatelet agents, including NSAIDs that cannot be stopped for surgery?
* Does the subject have a history of allergy or intolerance to flucytosine?
* Is the subject HIV positive?
* Does the subject have any gastrointestinal disease that would prevent him or her from being able to swallow or absorb flucytosine?
* Has the subject received any investigational treatment within the past 30 days?
* Is the subject breastfeeding?
* Does the patient have a history of prior malignancy, excluding basal or squamous cell carcinoma of the skin, with an expected survival of less than five years?

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2016-03-03 (Actual); Study Completion 2016-03-03 (Actual)

PRIMARY OUTCOMES:
Maximum feasible, safe, and tolerated dose of Toca 511 as measured by dose limiting toxicities. | 32 weeks

SECONDARY OUTCOMES:
Measure Toca 511 deposition in tumor at the time of resection by QT-PCR | At time of surgical resection
Measure how long Toca 511 stays in blood after IV administration by serum QT-PCR | 10 days
Safety and tolerability of Toca FC given at various doses and schedules as measured by dose limiting toxicities. | 32 weeks
Evaluate preliminary efficacy of Toca 511 and Toca FC by assessing overall survival, and tumor response rates. | Overall survival, Overall survival at 6 months (OS6), 9 months (OS9), and 12 months (OS12)
Evaluate preliminary efficacy by assessing landmark PFS [6 months] | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Asha Das, MD, Study Director — Tocagen Inc.; Steven Kalkanis, MD, Principal Investigator — Henry Ford Hospital
Locations (6):
- United States (6):
  - UC Irivine, Irvine, California
  - UCLA, Los Angeles, California
  - UC San Diego, Moores Cancer Center, San Diego, California
  - Henry Ford Hospital, Detroit, Michigan
  - JFK Medical Center New Jersery, Edison, New Jersey
  - Cleveland Clinic Foundation, Cleveland, Ohio

REFERENCES:
- [Background] Ostertag D, Amundson KK, Lopez Espinoza F, Martin B, Buckley T, Galvao da Silva AP, Lin AH, Valenta DT, Perez OD, Ibanez CE, Chen CI, Pettersson PL, Burnett R, Daublebsky V, Hlavaty J, Gunzburg W, Kasahara N, Gruber HE, Jolly DJ, Robbins JM. Brain tumor eradication and prolonged survival from intratumoral conversion of 5-fluorocytosine to 5-fluorouracil using a nonlytic retroviral replicating vector. Neuro Oncol. 2012 Feb;14(2):145-59. doi: 10.1093/neuonc/nor199. Epub 2011 Nov 9. PMID 22070930